CLINICAL TRIAL: NCT02513264
Title: Registry for Asthma Characterization and Recruitment 2 (ICAC-25)
Brief Title: Registry for Asthma Characterization and Recruitment 2
Acronym: RACR2
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Inner-City Asthma Consortium (Network)
Responsible Party: Sponsor
Other Study IDs: DAIT ICAC-25
Record Dates: First submitted 2015-07-23; First posted 2015-07-31 (Estimated); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Asthma
Keywords: Registry; Asthma; Inner City Asthma Consortium (ICAC) study eligibility
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Years
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: Yes

SUMMARY:
There is a need for people to take part in research studies to learn more about diseases and how to treat them. The Registry for Asthma Characterization and Recruitment 2 (RACR2) will create a database of participants with asthma and nasal allergies, or risk factors for these conditions, who are potentially eligible for future Inner City Asthma Consortium (ICAC) trials. The registry database will include assessments of various asthma and allergy characteristics to achieve a more efficient, selective recruitment of these participants for other protocols.

DETAILED DESCRIPTION:
The overall goal of the Registry for Asthma Characterization and Recruitment 2 (RACR2) is to create a database of participants who are potentially eligible for future Inner City Asthma Consortium (ICAC) clinical research studies. The registry will provide an avenue to assess various asthma and allergy characteristics, which will result in more efficient recruitment for current and future ICAC protocols.

Potential participants will be recruited via telephone or in person. Those deemed potentially eligible for a current protocol or protocol in development may be invited to the clinic for further data collection and assessments. This registry allows flexibility in selecting the eligibility criteria and data collection to match planned or upcoming ICAC protocols. At each stage of data collection, participants may be discontinued, put on hold, or invited to participate in further screening activities, depending on the likelihood that they will qualify for a future protocol. Participants may opt to withdraw their information or discontinue from the registry at any time, in person, by telephone, or in writing.

ELIGIBILITY:
Inclusion Criteria:

Eligibility criteria vary depending on recruitment needs for future ICAC protocols. Participants with asthma and participants without asthma, atopy, and rhinitis may be recruited at the same time or different times, depending on recruitment needs.

Certain characteristics or groups of characteristics within each criterion may be selected for periods of time across clinical sites or at each individually participating clinical site. For example, over a 6-month period, the Consortium could decide to recruit children aged 6 through 12 years with diagnosed asthma who have asthma symptoms, have a history of an asthma exacerbation, and reside in prespecified census tracts within the metropolitan statistical area. During selective recruitment periods, individuals who meet broader criteria may or may not be enrolled at the discretion of the Consortium.

1. All participants must resides within the metropolitan statistical area that includes the clinical site.
2. Participants with asthma are defined by having evidence of asthma. Evidence of asthma is defined by meeting at least one of the following criteria:

   * Clinician-diagnosed asthma
   * Asthma symptoms, history of an asthma exacerbation, or current use of asthma medication(s)
   * Recurrent wheezing
   * Wheezing apart from a cold

   At times of selective recruitment, participants with asthma may be required to meet more selective criteria above and may be required to meet one or more of the criteria in risk factors for asthma. Evidence of risk factors for asthma is defined by meeting at least one of the following criteria:
   * Parental history of asthma
   * Eczema or atopic dermatitis
   * Reported allergies to pets, food, indoor allergens, or outdoor allergens
   * Allergic sensitization by results of allergy skin testing or results of serum immunoglobulin E (IgE) testing
   * Rhinitis
3. Participants without asthma, atopy, and rhinitis must meet all of the following:

   * Negative history of an asthma diagnosis by a clinician
   * Negative history of a diagnosis of atopic dermatitis or eczema by a clinician
   * Negative history of a rhinitis diagnosis by a clinician
   * A forced expiratory volume at 1 second (FEV1) >= 5% predicted
   * Negative prick skin-tests to any of a panel of indoor and outdoor allergens
   * No current asthma as determined by the appropriate case report form
   * No current chronic rhinitis/sinusitis as determined by the appropriate case report form

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from enrollment:

1. Has any of the following chronic medical conditions: cardiac condition requiring daily medication, seizure disorder requiring daily medication, obvious severe mental retardation that prevents the participant from answering questions or following instructions, cystic fibrosis, immune deficiency, type 1 diabetes, allergic bronchopulmonary aspergillosis, or any other chronic medical condition at the discretion of the registry clinician
2. Does not primarily speak English (or Spanish at clinical sites with Spanish-speaking staff)
3. Has a primary caretaker who does not speak English (or Spanish at clinical sites with Spanish-speaking staff; not applicable if participant is able to provide consent)
4. Is a foster child (not applicable if participant is able to provide consent)
5. Is unwilling to sign the written informed consent form if of age, or parent/legal guardian is unwilling to sign the written informed consent if participant is not of age
6. Is unwilling to sign the assent form, if age appropriate

Participants who are pregnant will not be excluded or discontinued from RACR2 but will not undergo any procedures that are prohibited during pregnancy.

Ages: 1 Year to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Subjects who reside within the metropolitan statistical area of the clinical site and have clinician-diagnosed asthma, current symptoms of asthma, or risk factors for development of asthma. The population may at times include participants without asthma, atopy, and rhinitis.
Sampling Method: Non-Probability Sample
Enrollment: 1384 (Actual)
Dates: Start 2015-04-14; Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

PRIMARY OUTCOMES:
Number of participants with asthma and allergy characteristics | Year 7
  Characteristics of the participants enrolled in the registry will be assessed on a periodic basis (descriptive summary of diagnosis and parameters associated with the former).

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Pongracic, M.D., Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago; Edward M. Zoratti, M.D., Principal Investigator — Henry Ford Hospital
Locations (10):
- United States (10):
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Ann and Robert Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - St. Louis Children's Hospital, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - University of Texas Southwestern Medical School, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: National Institute of Allergy and Infectious Diseases — https://www.niaid.nih.gov
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — http://www.niaid.nih.gov/about/dait